CLINICAL TRIAL: NCT00781547
Title: Growth Hormone Treatment in Men With High Risk of Developing Type 2 Diabetes Mellitus
Acronym: GHDM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Gudmundur Johannsson, Department of Endocrinology, Sahlgrenska University Hospital, 413 45 Gothenburg, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GHNIDDM
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Abdominal Obesity; Metabolic Syndrome; Obesity
Keywords: growth hormone; obesity; abdominal obesity
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome; Obesity | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recombinant human growth hormone (Experimental): The subjects will receive treatment with recombinant human GH (Genotropin®) or placebo administered by a daily s.c. injection before bedtime. The initial dose of GH will be 0.4 IU per day increased to 0.8 IU after 2 weeks and to 1.2 IU after 4 weeks of treatment. Thus, the target dose is 1.2 IU per day which resembles approximately 0.015 IU/kg/day. The GH dose will be reduced by half in the event of side-effects
  Interventions: Drug: recombinant human growth hormone
- Placebo (Placebo Comparator)
  Interventions: Drug: recombinant human growth hormone

INTERVENTIONS:
Drug: recombinant human growth hormone — The subjects will receive treatment with recombinant human GH (Genotropin®) or placebo administered by a daily s.c. injection before bedtime. The initial dose of GH will be 0.4 IU per day increased to 0.8 IU after 2 weeks and to 1.2 IU after 4 weeks of treatment. Thus, the target dose is 1.2 IU per day which resembles approximately 0.015 IU/kg/day. The GH dose will be reduced by half in the event of side-effects

SUMMARY:
The overall aim of this study is to investigate the effects of GH treatment in men with the Metabolic Syndrome and a high risk of developing type 2 DM.

Forty men with abdominal obesity and impaired glucose tolerance will be randomized to two parallel treatment groups with GH and placebo for 12 months.

The subjects will receive treatment with recombinant human GH (Genotropin®) or placebo administered by a daily s.c. injection before bedtime. The initial dose of GH will be 0.4 IU per day increased to 0.8 IU after 2 weeks and to 1.2 IU after 4 weeks of treatment. Thus, the target dose is 1.2 IU per day which resembles approximately 0.015 IU/kg/day. The GH dose will be reduced by half in the event of side-effects. Oral and written instructions in terms of administration and dosage will be given.

The treatment can be discontinued by the patient. The treatment should be discontinued if malignancy is discovered, DM developes, if the subject experience a cerebrovascular disease and in the event of any other side-effects that is considered as serious.

The treatment code for each subject included in the trial will be kept at the Sahlgrenska University Hospital Pharmacy. This code can be broken on the request of the investigator.

Compliance will be assessed by collecting empty vials from the study subjects. The treatment is discontinued at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Fasting plasma glucose level ≥ 6.1 and ≤ 7.8 mmol/L (IFG) and/or a plasma glucose 2 hours after a 75g oral glucose load between 6.9-11.0 mmol/L (IGT).
* BMI > 25 kg/m2.
* Waist/hip ratio > 0.95

Exclusion Criteria:

* Proliferative diabetic retinopathy.
* Macro-albuminuri and/or serum creatinine >150mmol/L
* Known ischemic heart disease, previous stroke or claudicatio intermittence.
* Known malignancy.
* Other hormonal therapy.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1999-01; Primary Completion 2003-09 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | Baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
Fasting plasma glucose, serum insulin, HbA1c | Basline, 1,2,3,6,9 and 12 months
Sleep architecture | Baseline and 12 months
Visceral adipose tissue | Baseline and 12 months
Progress of atherosclerosis (IMT) | Baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum for Endocrinology and Metabolism, Sahlgenska University Hospital, Gothenburg, Sweden